CLINICAL TRIAL: NCT04178746
Title: PRONTO: Minimally Invasive Endoscopic Surgery Utilizing the Artemis Neuro Evacuation Device in Patients With Intraventricular Hemorrhage in the Hyper-Acute Phase
Brief Title: PRONTO: Artemis in the Removal of Intraventricular Hemorrhage in the Hyper-Acute Phase
Acronym: PRONTO
Status: Terminated | Type: Observational
Why Stopped: Business decision to focus on other studies. No safety concern.
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14087
Record Dates: First submitted 2019-10-28; First posted 2019-11-26 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Intracerebral Hemorrhage; Brain Hemorrhage; Intraventricular Hemorrhage
Keywords: intraventricular hemorrhage; IVH; stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- IVH subjects in the Hyper-Acute Phase: The purpose of this prospective, single center, single arm registry is to assess technical feasibility, peri-procedural complications, post-procedure imaging outcomes, and 30-day safety outcomes in approximately 20 subjects with intracerebral hemorrhages utilizing the Artemis Neuro Evacuation Device in the hyper-acute phase. For the purposes of this registry, the hyper-acute phase as defined by initiation of the MIS procedure no longer than 12 hours from initial NCCT scans and no longer than 18 hours since time patients last known well.
  Interventions: Device: Artemis Neuro Evacuation Device

INTERVENTIONS:
Device: Artemis Neuro Evacuation Device — The Artemis Neuro Evacuation Device is used for the controlled aspiration of tissue and/or fluid during surgery of the Ventricular System or Cerebrum in conjunction with a Penumbra Aspiration Pump.
  The Penumbra Aspiration Pump is indicated as a vacuum source for the Penumbra Aspiration Systems.
  The Artemis Device will be evaluated by descriptive statistics in this registry to assess its efficiency and reliability in minimally invasive, mechanical evacuation of hematoma in patients with intracranial hemorrhage under direct visualization and control using a neuroendoscope.

SUMMARY:
The purpose of this prospective, single center, single arm registry is to assess technical feasibility, peri-procedural complications, post-procedure imaging outcomes, and 30-day safety outcomes in subjects with intraventricular hemorrhages utilizing the Artemis Neuro Evacuation Device in the hyper-acute phase.

DETAILED DESCRIPTION:
The purpose of this prospective, single center, single arm registry is to assess technical feasibility, peri-procedural complications, post-procedure imaging outcomes, and 30-day safety outcomes in subjects with intracerebral hemorrhages utilizing the Artemis Neuro Evacuation Device in the hyper-acute phase.

The Artemis Neuro Evacuation Device is used for the controlled aspiration of tissue and/or fluid during surgery of the Ventricular System or Cerebrum in conjunction with a Penumbra Aspiration Pump.

The Penumbra Aspiration Pump is indicated as a vacuum source for the Penumbra Aspiration Systems.

The enrollment period will end once 20 evaluable subjects have been enrolled in the registry. Each subject will be in the registry for approximately 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years in age
2. Patients presenting with Intraventricular Hemorrhage (IVH) qualifying for hematoma evacuation
3. Controlled SBP ≤ 180 mmHg after initial NCCT scan and prior to the initiation of the MIS procedure
4. Hyper-acute phase, as defined by initiation of the MIS procedure no longer than 12 hours from initial NCCT scan and no longer than 18 hours since time patient last known well
5. Symptomatic with radiographic evidence of cerebral compression edema
6. Pre-stroke mRS 0 - 2

Exclusion Criteria:

1. Presence of tentorial herniation and/or Kernohan's phenomenon
2. Uncontrolled ICP as defined as > 25 mmHg for more than 30 min for 3 consecutive hours after External Ventricular Drain (EVD) placement
3. Requirement of insulin drip
4. Pregnancy or positive pregnancy test (either serum or urine). Women of child-bearing potential must have a negative pregnancy test prior to enrollment
5. Unable to obtain consent from patient or legally authorized representative (LAR) (for patients without competence)
6. Presenting epilepticus that is not controlled
7. Nonreversible coagulopathy (INR > 1.4) or platelet deficiency (< 75 x 103 cells/mm3) not able to be corrected with currently accepted treatment medications
8. Contraindication to conventional angiography, CTA, and MRA
9. Life expectancy of < 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spontaneous Intraventricular Hemorrhage not related to underlying vascular abnormality.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Efficacy Endpoint: Post-Procedural Hemorrhage reduction of ≥ 85% in hemorrhage volume assessed by CT at 24 hours | 24 hours
  Post-Procedural Hemorrhage reduction of ≥ 85% in hemorrhage volume assessed by CT at 24 hours
Safety Endpoint: Rate of mortality at 30 days | 30 days
  Rate of mortality at 30 days

SECONDARY OUTCOMES:
Time of admission at treating facility to discharge (Length of stay) | admission to discharge, a period of up to 30 days
Rate of Ventriculoperitoneal Shunt (VPS) placement within 30 days of procedure | 30 days
Procedure and device related SAEs | time of surgery up to 30-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Saphier, MD, Principal Investigator — Atlantic Neuroscience Institute
Locations (1):
- Atlantic Neuroscience Institute, Summit, New Jersey, United States